CLINICAL TRIAL: NCT00924638
Title: CRYptogenic STroke And underLying AF Trial
Brief Title: Study of Continuous Cardiac Monitoring to Assess Atrial Fibrillation After Cryptogenic Stroke
Acronym: CRYSTAL-AF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medtronic Cardiac Rhythm and Heart Failure (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: CRYSTAL-AF
Record Dates: First submitted 2009-06-17; First posted 2009-06-19 (Estimated); Results first posted 2014-07-28 (Estimated); Last update posted 2014-07-28 (Estimated); Status verified 2014-01

CONDITIONS: Cryptogenic Symptomatic Transient Ischemic Attack; Cryptogenic Ischemic Stroke
Keywords: atrial fibrillation; cryptogenic stroke; continuous monitoring; implantable loop recorder; insertable cardiac monitor
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Continuous Monitoring (Active Comparator): Continuous cardiac monitoring by the Reveal® XT Insertable Cardiac Monitor
  Interventions: Device: Reveal® XT Insertable Cardiac Monitor
- Control Arm (No Intervention): Follow-up at the same frequency, but with no Insertable Cardiac Monitor

INTERVENTIONS:
Device: Reveal® XT Insertable Cardiac Monitor — The Insertable Cardiac Monitor is implanted under the skin in the region of the thorax. It continuously monitors the heart's electrical activity for up to three years. ECG data are stored when the device detects a cardiac arrhythmia.
  Other Names: Reveal® XT
  Arms: Continuous Monitoring

SUMMARY:
The 2006 American Heart Association / American Stroke Association Council on Stroke Guidelines for Prevention of Stroke in Patients With Ischemic Stroke or Transient Ischemic recommended that patients with cryptogenic stroke take antithrombotic drugs (i.e. aspirin) in order to prevent a second stroke. When a stroke patient is found to have atrial fibrillation (AF), the guidelines recommend oral anticoagulation due to its superior efficacy over aspirin for stroke prevention. Physicians can best optimize the use of medicines only if they can precisely and correctly diagnose a patient's AF. The purpose of this study is to evaluate the time to first AF by 6 months' continuous rhythm monitoring versus control treatment in subjects with a recent cryptogenic stroke or Transient Ischemic Attack (TIA) without history of AF.

ELIGIBILITY:
Inclusion Criteria:

1. Recent cryptogenic symptomatic transient ischemic attack (TIA) or cryptogenic ischemic stroke.

Exclusion Criteria:

1. Known etiology of TIA or stroke.
2. Untreated hyperthyroidism.
3. Myocardial infarction less than 1 month prior to stroke or TIA.
4. Coronary bypass grafting less than 1 month prior to stroke or TIA.
5. Valvular disease requiring immediate surgical intervention.
6. History of AF or atrial flutter.
7. Patent Foramen Ovale (PFO) and PFO is or was an indication to start oral anticoagulation (OAC).
8. Permanent indication for OAC at enrollment.
9. Permanent contra-indication for OAC.
10. Included in another clinical trial.
11. Life expectancy less than 1 year.
12. Pregnant.
13. Indicated for Implantable Pulse Generator (IPG), Implantable Cardioverter-Defibrillator (ICD), Cardiac Resynchronization Therapy (CRT) or an implantable hemodynamic monitoring system.
14. Not fit, unable or unwilling to follow the required procedures of the protocol.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 447 (Actual)
Dates: Start 2009-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Brachmann, MD, Principal Investigator — Klinikum Coburg, Germany; Tommaso Sanna, MD, Principal Investigator — Catholic University, Italy; Hans Christoph Diener, MD, Principal Investigator — Klinik für Neurologie, Essen, Germany; Carlos Morillo, MD, Principal Investigator — McMaster Clinic, Hamilton, Ontario, Canada; Richard Bernstein, MD, PhD, Principal Investigator — Davee Department of Neurology, Chicago, IL USA; Vincenzo Di Lazzaro, MD, Principal Investigator — Catholic University Rome, Rome Italy; Rod Passman, MD, Principal Investigator — Northwestern Memorial Hospital, Chicago, IL USA; Marilyn Rymer, MD, Principal Investigator — St. Lukes Hospital of Kansas City, Kansas City, MI USA
Locations (55):
- United States (19):
  - El Camino Hospital, Mountain View, California
  - South Denver Cardiology / Swedish Medical Center, Denver, Colorado
  - Northwestern Memorial Hospital, Chicago, Illinois
  - Iowa Heart / Ruan Neurology, Des Moines, Iowa
  - Louisville Cardiology, Louisville, Kentucky
  - Cardiology Associates Research, LLC, Tupelo, Mississippi
  - Mid America Heart Institute / St. Lukes Hospital, Kansas City, Missouri
  - Washington University Medical School, St Louis, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Forsyth Medical Center, Winston-Salem, North Carolina
  - Ohio Health Research, Columbus, Ohio
  - Sacred Heart Medical Center, Eugene, Oregon
  - Central Bucks Specialists / Doylestown Hospital, Doylestown, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Lankenau, Wynnewood, Pennsylvania
  - Greenville Hospital System Cardiology/Cardiovascular Research, Greenville, South Carolina
  - St. Thomas Research Institute, Nashville, Tennessee
  - Baylor Research Institute, Dallas, Texas
  - University of Texas - Southwestern Medical Center, Dallas, Texas
- Austria (3):
  - LKH Universitätsklinikum Graz, Graz
  - AKH Linz, Linz
  - Landesklinikum Donauregion Tulln, Tulln
- Belgium (4):
  - UZ Antwerpen, Antwerp
  - Brussels Heart Center (St. Lean - St. Pierre), Brussels
  - UZ Leuven, Leuven
  - Cliniques Universitaires UCL Mont-Godinne, Mont Godinne
- Canada (2):
  - Hamilton Health Sciences / Hamilton General Hospital, Hamilton, Ontario
  - CHUS / Hopital Fleurimont, Sherbrooke, Quebec
- Skejby Hospital, Aarhus, Denmark
- Neurology clinic, Turku University Central Hospital, Turku, Finland
- France (3):
  - Hôpital Saint André -CHU de Bordeaux, Bordeaux
  - Clinique Parly II - Centre Hospitalier de Versailles, Le Chesnay
  - Hôpital de la Timone, Marseille
- Germany (10):
  - Klinikum Coburg GmbH, Coburg, Bavaria
  - Knappschaftskrankenhaus Bochum, Bochum
  - Klinikum Dortmund, Dortmund
  - Universitätsklinikum Essen, Essen
  - UMG, Goettingen, Göttingen
  - Universitätsklinikum der Ernst-Moritz-Arndt-Universität Greifswald, Greifswald
  - Asklepios Altona, Hamburg
  - Asklepios Barmbek, Hamburg
  - Städtisches Klinikum Karlsruhe GmbH, Karlsruhe
  - Kreiskrankenhaus Rastatt, Rastatt
- Henry Dunant General Hospital, Athens, Greece
- Italy (4):
  - Ospedale Misericordia di Grosseto, Grosseto
  - Ospedale di Imperia, Imperia
  - Policlinico Universitario Agostino Gemelli, Rome
  - Ospedale Bolognini, Seriate
- Netherlands (3):
  - Atrium Medisch Centrum, Heerlen
  - St. Antonius Ziekenhuis, Nieuwegein
  - UMC Utrecht, Utrecht
- Slovakia (2):
  - NUSCH, a.s. Bratislava, Bratislava
  - VUSCH Kosice, Košice
- Hospital Puerta de Hierro Majadahonda, Majadahonda, Spain
- University Hospital Lund, Lund, Sweden

REFERENCES:
- [Background] Sacco RL, Adams R, Albers G, Alberts MJ, Benavente O, Furie K, Goldstein LB, Gorelick P, Halperin J, Harbaugh R, Johnston SC, Katzan I, Kelly-Hayes M, Kenton EJ, Marks M, Schwamm LH, Tomsick T; American Heart Association; American Stroke Association Council on Stroke; Council on Cardiovascular Radiology and Intervention; American Academy of Neurology. Guidelines for prevention of stroke in patients with ischemic stroke or transient ischemic attack: a statement for healthcare professionals from the American Heart Association/American Stroke Association Council on Stroke: co-sponsored by the Council on Cardiovascular Radiology and Intervention: the American Academy of Neurology affirms the value of this guideline. Stroke. 2006 Feb;37(2):577-617. doi: 10.1161/01.STR.0000199147.30016.74. PMID 16432246
- [Background] Sinha AM, Diener HC, Morillo CA, Sanna T, Bernstein RA, Di Lazzaro V, Passman R, Beckers F, Brachmann J. Cryptogenic Stroke and underlying Atrial Fibrillation (CRYSTAL AF): design and rationale. Am Heart J. 2010 Jul;160(1):36-41.e1. doi: 10.1016/j.ahj.2010.03.032. PMID 20598970
- [Derived] Kaffenberger T, Bernhardt J, Koehler JL, Ziegler PD, Thijs VN. Ambulatory activity in stroke survivors associated with functional outcome and quality of life: An observational cohort study. Ann Phys Rehabil Med. 2022 Mar;65(2):101540. doi: 10.1016/j.rehab.2021.101540. Epub 2021 Nov 13. PMID 33984539
- [Derived] Witte KK, Tsivgoulis G, Reynolds MR, Tsintzos SI, Eggington S, Ismyrloglou E, Lyon J, Huynh M, Egea M, de Brouwer B, Ziegler PD, Franco N, Joglekar R, Rosemas SC, Liu S, Thijs V. Burden of oral anticoagulation in embolic stroke of undetermined source without atrial fibrillation. BMC Cardiovasc Disord. 2021 Mar 31;21(1):160. doi: 10.1186/s12872-021-01967-x. PMID 33789592
- [Derived] Verma N, Ziegler PD, Liu S, Passman RS. Incidence of atrial fibrillation among patients with an embolic stroke of undetermined source: Insights from insertable cardiac monitors. Int J Stroke. 2019 Feb;14(2):146-153. doi: 10.1177/1747493018798554. Epub 2018 Sep 10. PMID 30196791
- [Derived] Brachmann J, Morillo CA, Sanna T, Di Lazzaro V, Diener HC, Bernstein RA, Rymer M, Ziegler PD, Liu S, Passman RS. Uncovering Atrial Fibrillation Beyond Short-Term Monitoring in Cryptogenic Stroke Patients: Three-Year Results From the Cryptogenic Stroke and Underlying Atrial Fibrillation Trial. Circ Arrhythm Electrophysiol. 2016 Jan;9(1):e003333. doi: 10.1161/CIRCEP.115.003333. PMID 26763225
- [Derived] Bernstein RA, Di Lazzaro V, Rymer MM, Passman RS, Brachmann J, Morillo CA, Sanna T, Thijs V, Rogers T, Liu S, Ziegler PD, Diener HC. Infarct Topography and Detection of Atrial Fibrillation in Cryptogenic Stroke: Results from CRYSTAL AF. Cerebrovasc Dis. 2015;40(1-2):91-6. doi: 10.1159/000437018. Epub 2015 Jul 11. PMID 26182860
- [Derived] Sanna T, Diener HC, Passman RS, Di Lazzaro V, Bernstein RA, Morillo CA, Rymer MM, Thijs V, Rogers T, Beckers F, Lindborg K, Brachmann J; CRYSTAL AF Investigators. Cryptogenic stroke and underlying atrial fibrillation. N Engl J Med. 2014 Jun 26;370(26):2478-86. doi: 10.1056/NEJMoa1313600. PMID 24963567

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 447 subjects were enrolled in 55 study centers from 14 countries in North America and Europe, during the recruitment period of June 2009 to April 2012.
Pre-assignment Details: A total of 6 enrolled subjects were exited from the study prior to randomization due to: Eligibility criteria not met (n=4), and Subject withdrew consent (n=2).
Period: Overall Study
Arm/Group | Continuous Monitoring | Control Arm
Started | 221 (Randomized to Continuous Monitoring Arm) | 220 (Randomized to Control Arm)
Completed | 209 (Completed 6 months of follow-up) | 207 (Completed 6 months of follow-up)
Not Completed | 12 | 13
Not completed — Death | 3 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 5 | 7
Not completed — Physician Decision | 3 | 3

BASELINE CHARACTERISTICS:
Population: Intention-to-treat (ITT) population (all randomized subjects)
Groups:
- Total: Total of all reporting groups
Arm/Group | Continuous Monitoring | Control Arm | Total
Number analyzed (Participants) | 221 | 220 | 441
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (11.4) | 61.4 (11.3) | 61.5 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 82 | 161
  Male | 142 | 138 | 280
Region of Enrollment [Number; unit: participants]
  United States | 80 | 66 | 146
  Slovakia | 1 | 3 | 4
  Greece | 1 | 0 | 1
  Finland | 0 | 2 | 2
  Spain | 0 | 5 | 5
  Austria | 23 | 16 | 39
  Italy | 28 | 31 | 59
  France | 17 | 17 | 34
  Canada | 3 | 6 | 9
  Belgium | 14 | 27 | 41
  Denmark | 3 | 3 | 6
  Germany | 39 | 32 | 71
  Netherlands | 12 | 11 | 23
  Sweden | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: AF Detection Rate Within 6 Months
Description: Percentage of subjects with AF detected within 6 months of follow-up
Time Frame: 6 months
Population: Intention-to-treat (ITT) population (all randomized subjects)
Measure: Number; unit: percentage of participants
Arm/Group | Continuous Monitoring | Control Arm
Number analyzed (Participants) | 221 | 220
percentage of participants | 8.9 | 1.4
Statistical Analysis 1: Comparison: Continuous Monitoring vs Control Arm; Test type: Superiority or Other; p = 0.0006, Log Rank; Hazard Ratio (HR) = 6.4, 95% CI 2-sided [1.9 to 21.7] — A hazard ratio of > 1 indicates that Continuous Monitoring is superior to Control in detecting AF

2. Secondary Outcome: AF Detection Rate Within 12 Months
Description: Percentage of subjects with AF detected within 12 months of follow-up
Time Frame: 12 months
Population: Intention-to-treat (ITT) population (all randomized subjects)
Measure: Number; unit: percentage of participants
Arm/Group | Continuous Monitoring | Control Arm
Number analyzed (Participants) | 221 | 220
percentage of participants | 12.4 | 2.0
Statistical Analysis 1: Comparison: Continuous Monitoring vs Control Arm; Test type: Superiority or Other; p < 0.0001, Log Rank; Hazard Ratio (HR) = 7.3, 95% CI 2-sided [2.6 to 20.8] — A hazard ratio of > 1 indicates that Continuous Monitoring is superior to Control in detecting AF

3. Secondary Outcome: Incidence of Recurrent Stroke or TIA (Transient Ischemic Attack)
Description: Percentage of subjects with recurrent stroke or TIA within 12 months of follow-up
Time Frame: 12 months
Population: Intention-to-treat (ITT) population (all randomized subjects)
Measure: Number; unit: percentage of participants
Arm/Group | Continuous Monitoring | Control Arm
Number analyzed (Participants) | 221 | 220
percentage of participants | 7.1 | 9.1
Statistical Analysis 1: Comparison: Continuous Monitoring vs Control Arm; Test type: Superiority or Other; p = 0.25, Log Rank; Hazard Ratio (HR) = 0.68, 95% CI 2-sided [0.35 to 1.32] — A hazard ratio of < 1 indicates that the incidence rate of recurrent stroke or TIA is lower in the Continuous Monitoring arm compared to the Control arm

4. Secondary Outcome: Use of Oral Anticoagulation (OAC) Drugs
Description: Percentage of subjects who were using OAC drugs at the 12 months follow-up visit
Time Frame: 12 months
Population: Number of subjects who completed the 12-months follow-up visit
Measure: Number; unit: percentage of participants
Arm/Group | Continuous Monitoring | Control Arm
Number analyzed (Participants) | 197 | 185
percentage of participants | 14.7 | 6.0
Statistical Analysis 1: Comparison: Continuous Monitoring vs Control Arm; Test type: Superiority or Other; Mean Difference (Final Values) = 8.8, 95% CI 2-sided [2.8 to 14.8] — A difference of greater than 0 means that a higher percentage of subjects in the Continuous Monitoring arm were using the OAC drugs at the 12 months visit compared to the Control arm

5. Secondary Outcome: Use of Antiarrhythmic Drugs
Description: Percentage of subjects who were using antiarrhythmic drugs at the 12 months follow-up visit
Time Frame: 12 months
Population: Number of subjects who completed the 12 months follow-up visit
Measure: Number; unit: percentage of participants
Arm/Group | Continuous Monitoring | Control Arm
Number analyzed (Participants) | 197 | 185
percentage of participants | 2.0 | 1.6
Statistical Analysis 1: Comparison: Continuous Monitoring vs Control Arm; Test type: Superiority or Other; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-2.3 to 3.1] — A difference of greater than 0 means that a higher percentage of subjects in the Continuous Monitoring arm were using the anti-arrhythmic drugs at the 12 months visit compared to the Control arm

6. Secondary Outcome: Health Outcome as Evaluated by EQ-5D Questionnaire
Description: EQ-5D VAS (visual analog scale) quality of life score, which is a continuous measure of quality of life ranging from 0 (worst) to 100 (perfect health).
Time Frame: 12 months
Population: Number of subjects who reported EQ-5D VAS score at the 12 months visit
Measure: Mean (Standard Deviation); unit: units on a scale of 0 to 100
Arm/Group | Continuous Monitoring | Control Arm
Number analyzed (Participants) | 191 | 183
units on a scale of 0 to 100 | 78.9 (15.6) | 76.3 (16.2)
Statistical Analysis 1: Comparison: Continuous Monitoring vs Control Arm; Test type: Superiority or Other; p = 0.11, t-test, 2 sided

7. Secondary Outcome: Clinical Disease Burden and Care Pathway
Description: Incidence of cardiovascular (CV) or stroke/TIA related hospitalizations within 12 months
Time Frame: 12 months
Population: Intention-to-treat (ITT) population (all randomized subjects)
Measure: Number; unit: percentage of participants
Arm/Group | Continuous Monitoring | Control Arm
Number analyzed (Participants) | 221 | 220
percentage of participants | 10.5 | 7.2
Statistical Analysis 1: Comparison: Continuous Monitoring vs Control Arm; Test type: Superiority or Other; p = 0.33, Log Rank; Hazard Ratio (HR) = 1.37, 95% CI 2-sided [0.73 to 2.60] — A hazard ratio of < 1 indicates that the incidence rate of cardiovascular or stroke/TIA related hospitalization is lower in the Continuous Monitoring arm compared to the Control arm

8. Secondary Outcome: Impact of Patient Assistant Use on AF Diagnosis
Description: AF detection lag (days from AF occurrence to AF diagnosis) characterized by patient assistant (PA) use frequency
Time Frame: Follow-up closure
Population: Number of subjects in the Continuous Monitoring arm who had AF detected by the Insertable Cardiac Monitor (ICM) during the course of the study
Measure: Mean (Standard Deviation); unit: days from AF occurrence to AF diagnosis
Arm/Group | Continuous Monitoring
Number analyzed (Participants) | 39
days from AF occurrence to AF diagnosis
  PA used everyday | 14.0 (35.6)
  PA used most of the time (5-6 days/week) | 25.0 (31.4)
  PA used sometimes (3-4 days/week) | 174.8 (235.9)
  PA used rarely (1-2 days/week) | 15.3 (9.3)
  PA never used | 92.0 (NA) — Only one observation was available
  PA use frequency not reported | 20.0 (NA) — Only one observation was available

ADVERSE EVENTS:
Time Frame: Adverse events were collected throughout the study (from enrollment to exit). Average subject follow-up duration was 19.7 +/- 9.7 months (range: 0 - 42.7 months).
Description: Subjects were assessed for adverse events through scheduled follow-up visits at 6 month intervals, as well as through unscheduled visits as adverse events occur.
Arm/Group | Continuous Monitoring | Control Arm
Serious Adverse Events (participants affected / at risk) | 68/221 | 58/220
Other Adverse Events (participants affected / at risk) | 41/221 | 9/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Monitoring (N=221) | Control Arm (N=220)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Adnexa uteri mass (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Adverse drug reaction (General disorders) | 0 (0) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 6 (6) | 3 (3)
Atrial flutter (Cardiac disorders) | 2 (2) | 0 (0)
Atrial septal defect (Congenital, familial and genetic disorders) | 3 (3) | 5 (5)
Atrioventricular block second degree (Cardiac disorders) | 1 (1) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (2) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 11 (12) | 5 (5)
Cerebrovascular spasm (Nervous system disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 5 (5) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Chondrolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chondropathy (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Colonic polyp (Gastrointestinal disorders) | 2 (2) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (3) | 2 (2)
Coronary artery stenosis (Cardiac disorders) | 1 (1) | 0 (0)
Costochondritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Enteritis infectious (Infections and infestations) | 1 (1) | 0 (0)
Epilepsy (Nervous system disorders) | 1 (1) | 2 (2)
Face injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femoral arterial stenosis (Vascular disorders) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 1 (1)
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypertensive crisis (Vascular disorders) | 3 (3) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Implant site infection (Infections and infestations) | 3 (3) | 1 (1)
In-stent arterial restenosis (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Lung adenocarcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Macular degeneration (Eye disorders) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Medical device removal (Surgical and medical procedures) | 2 (2) | 0 (0)
Meniscal degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephropathy (Renal and urinary disorders) | 1 (1) | 0 (0)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0)
Peripheral vascular disorder (Vascular disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (3) | 2 (2)
Pocket erosion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Renal artery stenosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0)
Retinal artery embolism (Eye disorders) | 1 (1) | 0 (0)
Retinal artery occlusion (Eye disorders) | 2 (2) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Sick sinus syndrome (Cardiac disorders) | 3 (3) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 1 (1)
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Somatisation disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Sudden death (General disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Tachyarrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Tension headache (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 6 (6) | 9 (9)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1)
Urethral disorder (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Wolff-Parkinson-White syndrome (Cardiac disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Continuous Monitoring (N=221) | Control Arm (N=220)
Atrial fibrillation (Cardiac disorders) | 41 (60) | 9 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days